CLINICAL TRIAL: NCT02996851
Title: Traumatic Intracranial Hemorrhage in Users of Oral Antithrombotic Drugs: a Nationwide Pharmacoepidemiological Study
Brief Title: Traumatic Intracranial Hemorrhage in Users of Oral Antithrombotic Drugs
Status: Completed | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/958
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Intracranial Hemorrhage, Traumatic; Embolism and Thrombosis; Hematoma, Subdural, Intracranial
Keywords: Fibrinolytic Agents; Adverse effects; Norway; Registries
MeSH Terms: conditions — Intracranial Hemorrhage, Traumatic; Embolism and Thrombosis; Hematoma, Subdural, Intracranial

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Oral antithrombotic medications (OAM) are used for the prevention and treatment of thrombotic disorders. Among hemorrhagic complications of OAMs, intracranial hemorrhage (ICH) may have particularly devastating consequences with high morbidity, disability and mortality rates. The efficacy and safety profiles of OAMs are generally assessed in randomized controlled trials (RCT), but included patients are often highly selected and may not be representative of users in everyday clinical practice in terms of follow-up routines, age, gender, drug compliance, and polypharmacy. Moreover, it is often unclear whether or not traumatic ICHs are registered and reported in RCTs. Drifts in indications and treatment criteria may also be seen in everyday practice and drug discontinuation due to precautionary concerns including compliance, fall risk and comorbidity may be forgotten. Collectively, these factors may lead to other and potentially higher traumatic ICH rates in general clinical use than reported in RCTs.

The incidence rates of traumatic ICH in patients on OAMs in the general population remain unknown. In this nationwide registry based pharmacoepidemiological study we will investigate the incidence and case fatality of traumatic ICH in users of OAMs in Norway from 2008 through 2014.

ELIGIBILITY:
Inclusion Criteria:

* included in the Norwegian patient registry (NPR) and/or the Norwegian prescription database (NorPD)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (1) the Norwegian patient registry (NPR), which contains information about all admissions to Norwegian hospitals since 2008 with diagnoses coded according to the 10th revision of the International Classification of Diseases and (2) The Norwegian prescription database (NorPD), which contains information about all prescriptions dispensed in Norway since 2004 including type of drug according to the Anatomical Therapeutic Chemical (ATC) classification system, number of Defined Daily Doses (DDD) as defined by the World Health Organization, date of dispensing, quantity dispensed, and drug strength and formulation. The National Registry provides information to NPR and NorPD on vital status (dead or alive).
Sampling Method: Non-Probability Sample
Enrollment: 6279 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
incidence of intracranial hemorrhage requiring hospital admission | at least 12 months following intracranial hemorrhage
  Age- and gender-adjusted comparisons of annual incidence rates will be carried out

SECONDARY OUTCOMES:
incidence of fatal traumatic intercranial hemorrhage defined as death within 90 days of admission | 90 days
  Age- and gender-adjusted comparisons of annual incidence rates will be carried out.
overall survival following traumatic intracranial hemorrhage | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Gulati, md phd, Principal Investigator — Norwegian University of Science and Technology

IPD SHARING:
Plan to Share IPD: No